CLINICAL TRIAL: NCT00530374
Title: Impact of Oral Iron Supplementation With Sprinkles on Infectious Morbidity When Moderate to Severe Pediatric Malnutrition Is Highly Prevalent - A Non-Inferiority Safety Trial
Brief Title: Impact of Sprinkles on Infectious Morbidity When Moderate to Severe Pediatric Malnutrition Is Highly Prevalent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Bangladesh Rural Advancement Committee (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Stanley Zlotkin, Chief, Global Child Health, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000009576
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Malnutrition; Iron Deficiency
Keywords: Pediatrics; Malnutrition; Iron Deficiency; Sprinkles; Oral Iron Supplementation
MeSH Terms: conditions — Malnutrition; Iron Deficiencies | interventions — Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Each child in this group will receive daily supplementation of Iron Sprinkles with a single sachet for 60 days
  Interventions: Dietary Supplement: Oral Iron Supplement
- 2 (Placebo Comparator): Each child in this group will receive daily supplementation of placebo Sprinkles with a single sachet for 60 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral Iron Supplement — Iron Sprinkles are provided as a powder in a single-dose sachet to be taken once daily for 60 days
  Other Names: Sprinkles
  Arms: 1
Dietary Supplement: Placebo — Placebo Sprinkles are provided as a powder in a single-dose sachet to be taken once daily for 60 days
  Other Names: Placebo Sprinkles
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety profile of oral iron supplementation (OIS) with Sprinkles in a pediatric population with high prevalence of Iron deficiency (ID) and moderate or severe malnutrition (MSM); the efficacy profile will also be investigated.

DETAILED DESCRIPTION:
Iron deficiency (ID) affects many children in developing countries. Anemia and impaired brain development are its most significant consequences. These may be prevented by giving oral iron supplements (OIS), such as Sprinkles. ID treatment was controversial because high dose parenteral iron therapy is strongly associated with severe infections when given to severely malnourished children. Many studies have since demonstrated the safety of low dose OIS. WHO guidelines reflect this finding: population-wide iron supplementation campaign (PWISC), without prior screening, is recommended when ID prevalence is ≥ 40%.

However, a gap in the safety evidence has been identified: children with moderate or severe malnutrition (MSM) are strikingly absent from the studies performed to date to investigate the link between OIS and infectious morbidities. In this context, PWISC may have unrecognized deleterious effects when the prevalence of MSM is high, since safety is assumed, but incorrectly extrapolated from available evidence.

We wish to emphasize an additional concern with regards to safety studies published thus far: all were designed as superiority trials. In this context, it is statistically incorrect to conclude that failure to show a significant difference between iron and placebo means that their respective side-effect profiles are similar.

ELIGIBILITY:
Inclusion Criteria:

* children aged 12 - 24 months
* moderate to severe malnutrition (MSM), defined as weight-for-age Z-score ≤ -2 based on the National Center for Health Statistics (NCHS) standards

Exclusion Criteria:

* severe anemia (hemoglobin ≤70g/L)
* near normal hemoglobin concentration (>100g/L)
* weight-for-height <-3 z-score (severe wasting)
* kwashiorkor (defined as evidence of edema)
* congenital abnormality or disease
* treatment with iron supplements in the past 3 months
* inclusion in a nutrition program in the past
* chronic illness other than malnutrition.

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 268 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
A composite score based on the sum of all distinct episodes of diarrhea, dysentery and lower respiratory tract infections | 2 distinct and consecutive phases of 6 months each

SECONDARY OUTCOMES:
Incidence of death and fever without a source [Safety] | 2 distinct and consecutive phases of 6 months each
Change in haemoglobin concentration after Sprinkles supplementation [Efficacy] | 2 distinct and consecutive phases of 6 months each

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Zlotkin, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- Village of Shombhuganj, Shombhuganj, Mymensingh District, Bangladesh

REFERENCES:
- [Derived] Lemaire M, Islam QS, Shen H, Khan MA, Parveen M, Abedin F, Haseen F, Hyder Z, Cook RJ, Zlotkin SH. Iron-containing micronutrient powder provided to children with moderate-to-severe malnutrition increases hemoglobin concentrations but not the risk of infectious morbidity: a randomized, double-blind, placebo-controlled, noninferiority safety trial. Am J Clin Nutr. 2011 Aug;94(2):585-93. doi: 10.3945/ajcn.110.009316. Epub 2011 Jun 29. PMID 21715512